CLINICAL TRIAL: NCT03607487
Title: A Phase 2, Dose-Escalation, Placebo-Controlled Study of the Safety of INCB054707 in Participants With Hidradenitis Suppurativa
Brief Title: A Placebo-Controlled Study of the Safety of INCB054707 in Participants With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 54707-203; 2018-000827-15 (EudraCT Number)
Record Dates: First submitted 2018-06-25; First posted 2018-07-31 (Actual); Results first posted 2020-09-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; Janus kinase (JAK) inhibitor; skin disease
MeSH Terms: conditions — Hidradenitis Suppurativa; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): INCB054707 at the Cohort 1 dose or placebo.
  Interventions: Drug: INCB054707; Drug: Placebo
- Cohort 2 (Experimental): INCB054707 at the Cohort 2 dose or placebo.
  Interventions: Drug: INCB054707; Drug: Placebo
- Cohort 3 (Experimental): INCB054707 at the Cohort 3 dose or placebo.
  Interventions: Drug: INCB054707; Drug: Placebo

INTERVENTIONS:
Drug: INCB054707 — INCB054707 tablet administered orally once daily at the protocol-defined dose.
  Other Names: Povorcitinib
Drug: Placebo — Placebo tablet administered orally once daily.

SUMMARY:
The purpose of this study is to evaluate the safety of INCB054707 over an 8-week treatment period in men and women with moderate to severe hidradenitis suppurativa.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS (confirmed by a dermatologist) with a disease duration of at least 6 months before screening.
* Stable course of HS for at least 90 days before screening, as determined by the investigator.
* HS lesions present in at least 2 distinct anatomic areas, 1 of which must be Hurley Stage II or Hurley Stage III at screening.
* Total AN count of at least 3 at screening and baseline.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Women who are currently pregnant or lactating.
* Presence of > 20 draining fistulas at screening and baseline.
* Participants with protocol-defined concurrent conditions or history of other diseases.
* Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF), defined as ≥ 450 msec.
* Positive test result for tuberculosis from the QuantiFERON-TB Gold test, or T-SPOT.TB test at screening.
* A history of active tuberculosis (treated or untreated) or a history of untreated latent tuberculosis.
* Positive serology test results for HIV, hepatitis B surface antigen, hepatitis B virus core antibody, or hepatitis C virus (HCV antibody with positive HCV-RNA) at screening.
* Decreased blood cell counts at screening per protocol-defined criteria.
* Severely impaired liver function (Child-Pugh Class C) or alanine aminotransferase or aspartate aminotransferase levels ≥ 1.5 × upper limit of normal at screening.
* Impaired renal function with serum creatinine > 1.5 mg/dL at screening.
* Use of protocol-prohibited medications.
* Known or suspected allergy to INCB054707 or any component of the study drug.
* Known history of clinically significant drug or alcohol abuse in the last year before baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation
Locations (13):
- Canada (9):
  - Investigative Site, Winnipeg, Manitoba
  - Investigative Site, Fredericton, New Brunswick
  - Investigative Site, Barrie, Ontario
  - Investigative Site, London, Ontario
  - Investigative Site 009, Markham, Ontario
  - Investigative Site 008, Richmond Hill, Ontario
  - Investigative Site 007, Windsor, Ontario
  - Investigative Site, Drummondville, Quebec
  - Investigative Site, Saint-Jérôme, Quebec
- Denmark (2):
  - Investigative Site, Aarhus
  - Investigative Site, Roskilde
- Germany (2):
  - Investigative Site, Bochum, Noth Rhine-Westphalia
  - Investigative Site, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alavi A, Hamzavi I, Brown K, Santos LL, Zhu Z, Liu H, Howell MD, Kirby JS. Janus kinase 1 inhibitor INCB054707 for patients with moderate-to-severe hidradenitis suppurativa: results from two phase II studies. Br J Dermatol. 2022 May;186(5):803-813. doi: 10.1111/bjd.20969. Epub 2022 Mar 6. PMID 34978076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 different sites in Canada, 2 different sites in Germany and 1 site in Denmark
Pre-assignment Details: A total of 43 participants were screened for enrollment in the study, 8 did not meet the eligibility criteria. A total of 35 participants were randomized to one of the treatment groups.
Groups:
- Placebo: Placebo was administered QD over an 8 week treatment period.
- INCB054707 at 30 mg: INCB054707 was administered at 30 mg QD over an 8 week treatment period.
- INCB054707 at 60 mg: INCB054707 was administered at 60 mg QD over an 8 week treatment period.
- INCB054707 at 90 mg: INCB054707 was administered at 90 mg QD over an 8 week treatment period.
Period: Overall Study
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Started | 9 | 9 | 9 | 8
Completed | 7 | 9 | 9 | 7
Not Completed | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg | Total
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (16.70) | 41.0 (11.53) | 42.2 (11.96) | 42.8 (14.62) | 41.5 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 8 | 5 | 28
  Male | 1 | 2 | 1 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 8 | 7 | 9 | 7 | 31
  Black/African-American | 0 | 0 | 0 | 1 | 1
  American-Indian/Alaska Native | 0 | 2 | 0 | 0 | 2
  Other | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 7 | 9 | 8 | 33
  Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Apparent Oral Clearance of INCB054707
Description: To determine the systemic exposure to INCB054707. Dependent upon the final compartmental model describing INCB054707.
Time Frame: Predose Day 1, Week 4, and 8, Postdose Day1, week 2,4,6, and 8
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Mean (Standard Deviation); unit: L/hr
Groups:
- INCB54707: INCB54707 was administered at either 30,60, or 90 mg. All samples from different dose groups were combined for this analysis.
Arm/Group | INCB54707
Number analyzed (Participants) | 26
L/hr | 5.27 (2.89)

2. Secondary Outcome: Apparent Oral Volume of Distribution of INCB054707
Description: To determine the systemic exposure to INCB054707. Dependent upon the final compartmental model describing INCB054707.
Time Frame: Predose Day 1, Week 4, and 8, Postdose Day1, week 2,4,6, and 8
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Mean (Standard Deviation); unit: L
Arm/Group | INCB54707
Number analyzed (Participants) | 26
L | 239 (85.7)

3. Secondary Outcome: Proportion of Participants Achieving a Hidradenitis Suppurativa Clinical Response (HiSCR) at Each Visit
Description: HiSCR defined as at least 50% reduction in abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to baseline.
Time Frame: Weeks 1, 2, 4, 6, 8, Early Termination and Follow-up (Up to 3 months)
Population: Full Analysis Set Population. Full Analysis Set Population In placebo group 1 participant discontinued the study before week 1, second participant missed all the visits and only had early termination visit. In the 90mg group 1 participant missed week 1 visit and a second participant discontinued before the follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Participants
  Week 1: number analyzed (Participants) | 7 | 9 | 9 | 7
  Week 1: Yes | 1 | 1 | 4 | 2
  Week 1: No | 6 | 8 | 5 | 5
  Week 2: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 2: Yes | 1 | 6 | 5 | 4
  Week 2: No | 6 | 3 | 4 | 4
  Week 4: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 4: Yes | 3 | 5 | 5 | 5
  Week 4: No | 4 | 4 | 4 | 3
  Week 6: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 6: Yes | 3 | 3 | 6 | 6
  Week 6: No | 4 | 6 | 3 | 2
  Week 8: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 8: Yes | 4 | 5 | 5 | 7
  Week 8: No | 3 | 4 | 4 | 1
  Follow Up: number analyzed (Participants) | 7 | 9 | 9 | 7
  Follow Up: Yes | 3 | 3 | 1 | 4
  Follow Up: No | 4 | 6 | 8 | 3
  Early Termination: number analyzed (Participants) | 1 | 0 | 0 | 0
  Early Termination: Yes | 0 | 0 | 0 | 0
  Early Termination: No | 1 | 0 | 0 | 0

4. Secondary Outcome: Proportion of Participants Achieving an AN Count of 0 to 2 at Each Visit
Description: AN defined as abscess and inflammatory nodule count.
Time Frame: Baseline,Weeks 1, 2, 4, 6, 8, Early Termination and Follow-up (Up to 3 months)
Population: Full Analysis Set Population In placebo group 1 participant discontinued the study before week 1, second participant missed all the visits and only had early termination visit. In the 90mg group 1 participant missed week 1 visit and a second participant discontinued before the follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Participants
  Baseline: Yes | 0 | 0 | 0 | 1
  Baseline: No | 9 | 9 | 9 | 7
  Week 1: number analyzed (Participants) | 7 | 9 | 9 | 7
  Week 1: Yes | 0 | 0 | 2 | 2
  Week 1: No | 7 | 9 | 7 | 5
  Week 2: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 2: Yes | 0 | 3 | 5 | 4
  Week 2: No | 7 | 6 | 4 | 4
  Week 4: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 4: Yes | 2 | 3 | 6 | 5
  Week 4: No | 5 | 6 | 3 | 3
  Week 6: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 6: Yes | 3 | 2 | 5 | 5
  Week 6: No | 4 | 7 | 4 | 3
  Week 8: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 8: Yes | 4 | 4 | 4 | 5
  Week 8: No | 3 | 5 | 5 | 3
  Follow Up: number analyzed (Participants) | 7 | 9 | 9 | 7
  Follow Up: Yes | 1 | 3 | 0 | 4
  Follow Up: No | 6 | 6 | 9 | 3
  Early Termination: number analyzed (Participants) | 1 | 0 | 0 | 0
  Early Termination: Yes | 0 | 0 | 0 | 0
  Early Termination: No | 1 | 0 | 0 | 0

5. Secondary Outcome: Mean Change From Baseline in the Hidradenitis Suppurativa Pain Numeric Rating Scale (HS Pain NRS) Scores at Each Visit
Description: An 11-point scale used to assess the worst skin pain and the average skin pain due to HS. Skin pain ranges from 0 ("no skin pain") to 10 ("skin pain as bad as you can imagine").
Time Frame: Baseline,Weeks 1, 2, 4, 6, 8, Early Termination and Follow-up (Up to 3 months)
Population: Full Analysis Set Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Units on a scale
  Mean change from Baseline to Week 1: number analyzed (Participants) | 6 | 5 | 8 | 6
  Mean change from Baseline to Week 1 | 0.2 (1.39) | -0.8 (1.13) | -0.3 (1.06) | -1.5 (1.04)
  Mean change from Baseline to Week 2: number analyzed (Participants) | 6 | 5 | 8 | 7
  Mean change from Baseline to Week 2 | -0.1 (1.49) | -1.5 (1.18) | -1.1 (0.91) | -3.3 (3.06)
  Mean change from Baseline to Week 4: number analyzed (Participants) | 6 | 5 | 8 | 7
  Mean change from Baseline to Week 4 | -0.3 (2.09) | -2.0 (2.02) | -1.4 (1.56) | -3.6 (3.30)
  Mean change from Baseline to Week 6: number analyzed (Participants) | 6 | 4 | 8 | 7
  Mean change from Baseline to Week 6 | 0.0 (3.49) | -0.9 (0.90) | -2.0 (1.55) | -3.4 (3.05)
  Mean change from Baseline to Week 8: number analyzed (Participants) | 6 | 4 | 8 | 7
  Mean change from Baseline to Week 8 | 0.3 (2.77) | -2.2 (2.18) | -1.4 (1.44) | -3.1 (3.28)
  Mean change from Baseline to Follow Up: number analyzed (Participants) | 3 | 3 | 8 | 4
  Mean change from Baseline to Follow Up | 2.6 (2.62) | -2.7 (2.20) | -0.8 (0.97) | -1.2 (1.91)

6. Secondary Outcome: Mean Change From Baseline in the Modified Sartorius Scale Score
Description: The Sartorius Scale is used to quantify the severity of HS. Points are awarded for 12 body areas (left and right axillae, left and right sub/inframammary areas, intermammary area, left and right buttocks, left and right inguino-crural folds, perianal area, perineal area, and other). For each area, points are awarded for nodules (2 points for each); abscesses (4 points); fistulas (4 points); scars (1 point); longest distance between two lesions (2-6 points, 0 if no lesions); and if lesions are separated buy normal skin (yes-0 point; no-6 points). The total Sartorius Scale score is the sum of the 12 regional scores. Scale scores range from 0 to infinite, with larger scores representing higher severity of HS.
Time Frame: From baseline up to week 8
Population: Full Analysis Set Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Units on a scale | -36.4 (35.83) | -41.9 (36.84) | -59.2 (48.48) | -54.6 (55.42)

7. Secondary Outcome: Mean Change From Baseline in the Number of Draining Fistulas Count at Each Visit.
Description: Defined as fistulas that drain serous or purulent fluid, either spontaneously or by gentle palpation.
Time Frame: Baseline,Weeks 1, 2, 4, 6, 8 and Follow-up (Up to 3 months)
Population: Full Analysis Set Population
Measure: Mean (Standard Deviation); unit: Number of Fistulas
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Number of Fistulas
  Week 1: number analyzed (Participants) | 7 | 9 | 9 | 7
  Week 1 | -0.1 (0.38) | -0.1 (1.27) | -0.8 (2.39) | -0.3 (0.49)
  Week 2: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 2 | 0.0 (1.53) | -0.9 (1.05) | -2.1 (3.48) | -0.8 (2.19)
  Week 4: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 4 | -0.9 (2.79) | -0.6 (1.01) | -2.0 (3.57) | -0.9 (2.53)
  Week 6: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 6 | -1.3 (2.69) | -0.4 (1.74) | -2.1 (3.30) | -0.6 (2.72)
  Week 8: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 8 | -1.0 (3.06) | -0.3 (1.66) | -2.0 (3.35) | -0.6 (3.85)
  Follow Up: number analyzed (Participants) | 7 | 9 | 9 | 7
  Follow Up | -0.4 (3.10) | 0.1 (1.69) | -2.2 (3.19) | -1.3 (3.86)

8. Secondary Outcome: Proportion of Participants at Each Category of Hurley Stage
Description: The Hurley classification is a static score and was originally designed for selection of the appropriate treatment modality in a certain body region. The assessor determines the Hurley stage in each affected anatomical region. If more than 1 stage is present in the same region, the worst stage in that region is documented. The participant will be assigned an overall Hurley stage classification corresponding to the stage of the worst involved anatomical region. The definition of each Hurley stage is as follows:
  Stage I : Abscess formation, single or multiple, without sinus tracts and cicatrization (scarring).
  Stage II : One or more widely separated recurrent abscesses with tract formation and cicatrization (scarring).
  Stage III : Multiple interconnected tracts and abscesses across the entire area, with diffuse or near diffuse involvement.
Time Frame: Baseline and Week 8
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Participants
  Baseline: Stage I | 0 | 0 | 0 | 0
  Baseline: Stage II | 4 | 9 | 5 | 7
  Baseline: Stage III | 5 | 0 | 4 | 1
  Baseline: No HS | 0 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 8: Stage I | 1 | 3 | 3 | 0
  Week 8: Stage II | 3 | 6 | 5 | 7
  Week 8: Stage III | 3 | 0 | 0 | 0
  Week 8: No HS | 0 | 0 | 1 | 1

9. Secondary Outcome: Proportions of Participants in Each HS Patient Global Impression of Change (PGIC) Category During the Treatment Period
Description: The HS-PGIC consists of 1 self-administered item that assesses change in the severity of skin in the HS area. The participant will answer the following: Since your last visit, your HS is: (1) very much improved, (2) much improved, (3) minimally improved, (4) no change, (5) minimally worse, (6) much worse, or (7) very much worse.
Time Frame: Up to 12 weeks
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Participants
  Week 1: number analyzed (Participants) | 7 | 9 | 9 | 7
  Week 1: 1 | 0 | 0 | 0 | 0
  Week 1: 2 | 0 | 1 | 0 | 0
  Week 1: 3 | 0 | 3 | 3 | 3
  Week 1: 4 | 4 | 2 | 4 | 2
  Week 1: 5 | 3 | 3 | 1 | 2
  Week 1: 6 | 0 | 0 | 1 | 0
  Week 1: 7 | 0 | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 2: 1 | 0 | 1 | 0 | 0
  Week 2: 2 | 0 | 1 | 2 | 3
  Week 2: 3 | 3 | 4 | 3 | 1
  Week 2: 4 | 1 | 2 | 3 | 3
  Week 2: 5 | 3 | 1 | 1 | 1
  Week 2: 6 | 0 | 0 | 0 | 0
  Week 2: 7 | 0 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 4: 1 | 0 | 1 | 2 | 0
  Week 4: 2 | 0 | 1 | 1 | 3
  Week 4: 3 | 3 | 2 | 1 | 1
  Week 4: 4 | 2 | 2 | 2 | 2
  Week 4: 5 | 2 | 1 | 2 | 2
  Week 4: 6 | 0 | 1 | 1 | 0
  Week 4: 7 | 0 | 1 | 0 | 0
  Week 6: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 6: 1 | 0 | 0 | 1 | 0
  Week 6: 2 | 1 | 1 | 1 | 2
  Week 6: 3 | 3 | 2 | 3 | 2
  Week 6: 4 | 1 | 4 | 1 | 4
  Week 6: 5 | 2 | 1 | 3 | 0
  Week 6: 6 | 0 | 1 | 0 | 0
  Week 6: 7 | 0 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 8: 1 | 0 | 0 | 0 | 1
  Week 8: 2 | 0 | 3 | 1 | 0
  Week 8: 3 | 1 | 1 | 3 | 1
  Week 8: 4 | 5 | 3 | 4 | 2
  Week 8: 5 | 1 | 1 | 1 | 3
  Week 8: 6 | 0 | 1 | 0 | 1
  Week 8: 7 | 0 | 0 | 0 | 0
  Early Termination: number analyzed (Participants) | 1 | 0 | 0 | 0
  Early Termination: 1 | 0 | 0 | 0 | 0
  Early Termination: 2 | 0 | 0 | 0 | 0
  Early Termination: 3 | 0 | 0 | 0 | 0
  Early Termination: 4 | 1 | 0 | 0 | 0
  Early Termination: 5 | 0 | 0 | 0 | 0
  Early Termination: 6 | 0 | 0 | 0 | 0
  Early Termination: 7 | 0 | 0 | 0 | 0
  Follow Up: number analyzed (Participants) | 7 | 9 | 9 | 7
  Follow Up: 1 | 0 | 0 | 0 | 0
  Follow Up: 2 | 0 | 1 | 0 | 0
  Follow Up: 3 | 1 | 1 | 0 | 0
  Follow Up: 4 | 1 | 2 | 2 | 1
  Follow Up: 5 | 3 | 2 | 2 | 3
  Follow Up: 6 | 2 | 3 | 4 | 0
  Follow Up: 7 | 0 | 0 | 1 | 3

10. Secondary Outcome: Actual Measurements in HS-PGIC at Each Visit
Description: as for outcome 9
Time Frame: Up to 12 weeks
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Participants
  Week 1: number analyzed (Participants) | 7 | 9 | 9 | 7
  Week 1: 1 | 0 | 0 | 0 | 0
  Week 1: 2 | 0 | 1 | 0 | 0
  Week 1: 3 | 0 | 3 | 3 | 3
  Week 1: 4 | 4 | 2 | 4 | 2
  Week 1: 5 | 3 | 3 | 1 | 2
  Week 1: 6 | 0 | 0 | 1 | 0
  Week 1: 7 | 0 | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 2: 1 | 0 | 1 | 0 | 0
  Week 2: 2 | 0 | 1 | 2 | 3
  Week 2: 3 | 3 | 4 | 3 | 1
  Week 2: 4 | 1 | 2 | 3 | 3
  Week 2: 5 | 3 | 1 | 1 | 1
  Week 2: 6 | 0 | 0 | 0 | 0
  Week 2: 7 | 0 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 4: 1 | 0 | 1 | 2 | 0
  Week 4: 2 | 0 | 1 | 1 | 3
  Week 4: 3 | 3 | 2 | 1 | 1
  Week 4: 4 | 2 | 2 | 2 | 2
  Week 4: 5 | 2 | 1 | 2 | 2
  Week 4: 6 | 0 | 1 | 1 | 0
  Week 4: 7 | 0 | 1 | 0 | 0
  Week 6: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 6: 1 | 0 | 0 | 1 | 0
  Week 6: 2 | 1 | 1 | 1 | 2
  Week 6: 3 | 3 | 2 | 3 | 2
  Week 6: 4 | 1 | 4 | 1 | 4
  Week 6: 5 | 2 | 1 | 3 | 0
  Week 6: 6 | 0 | 1 | 0 | 0
  Week 6: 7 | 0 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 7 | 9 | 9 | 8
  Week 8: 1 | 0 | 0 | 0 | 1
  Week 8: 2 | 0 | 3 | 1 | 0
  Week 8: 3 | 1 | 1 | 3 | 1
  Week 8: 4 | 5 | 3 | 4 | 2
  Week 8: 5 | 1 | 1 | 1 | 3
  Week 8: 6 | 0 | 1 | 0 | 1
  Week 8: 7 | 0 | 0 | 0 | 0
  Early Termination: number analyzed (Participants) | 1 | 0 | 0 | 0
  Early Termination: 1 | 0 | 0 | 0 | 0
  Early Termination: 2 | 0 | 0 | 0 | 0
  Early Termination: 3 | 0 | 0 | 0 | 0
  Early Termination: 4 | 1 | 0 | 0 | 0
  Early Termination: 5 | 0 | 0 | 0 | 0
  Early Termination: 6 | 0 | 0 | 0 | 0
  Early Termination: 7 | 0 | 0 | 0 | 0
  Follow Up: number analyzed (Participants) | 7 | 9 | 9 | 7
  Follow Up: 1 | 0 | 0 | 0 | 0
  Follow Up: 2 | 0 | 1 | 0 | 0
  Follow Up: 3 | 1 | 1 | 0 | 0
  Follow Up: 4 | 1 | 2 | 2 | 1
  Follow Up: 5 | 3 | 2 | 2 | 3
  Follow Up: 6 | 2 | 3 | 4 | 0
  Follow Up: 7 | 0 | 0 | 1 | 3

11. Secondary Outcome: Proportion of Participants With Change From Baseline Hurley Stage
Description: as for outcome 8
Time Frame: Baseline and Week 8
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Participants
  Baseline: Stage I | 0 | 0 | 0 | 0
  Baseline: Stage II | 4 | 9 | 5 | 7
  Baseline: Stage III | 5 | 0 | 4 | 1
  Baseline: No HS | 0 | 0 | 0 | 0
  Baseline: Missing | 0 | 0 | 0 | 0
  Week 8: Stage I | 1 | 3 | 3 | 0
  Week 8: Stage II | 3 | 6 | 5 | 7
  Week 8: Stage III | 3 | 0 | 0 | 0
  Week 8: No HS | 0 | 0 | 1 | 1
  Week 8: Missing | 2 | 0 | 0 | 0

12. Primary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: TEAE is defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug. Grading was performed using guidance from the CTCAE v 4.03. A grade 3 and above would constitute as "severe".
Time Frame: Up to 12 weeks
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg
Number analyzed (Participants) | 9 | 9 | 9 | 8
Participants
  Grade 1 | 2 | 6 | 4 | 1
  Grade 2 | 2 | 2 | 2 | 3
  Grade 3 | 0 | 0 | 0 | 3
  Grade 4 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Groups:
- Total: Total
Arm/Group | Placebo | INCB054707 at 30 mg | INCB054707 at 60 mg | INCB054707 at 90 mg | Total
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/8 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/8 | 0/35
Other Adverse Events (participants affected / at risk) | 4/9 | 8/9 | 6/9 | 7/8 | 25/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | INCB054707 at 30 mg (N=9) | INCB054707 at 60 mg (N=9) | INCB054707 at 90 mg (N=8) | Total (N=35)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acne cystic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 7 (7)
Folliculitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3) | 2 (4) | 6 (9)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT03607487/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03607487/SAP_001.pdf